CLINICAL TRIAL: NCT07151703
Title: Carrier-Assisted Topical Application Versus Intranasal Injection of Autologous Platelet-Rich Plasma for Olfactory Dysfunction: A Randomized Controlled Trial
Brief Title: Topical Versus Injection PRP for Olfactory Dysfunction
Acronym: TOP-IN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yun-Ting Chao, Dr., Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-06-010C; after funding being approved (Other Grant/Funding Number: Taipei Veterans General Hospital)
Record Dates: First submitted 2025-08-16; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Olfactory Dysfunction; Anosmia; Hyposmia
Keywords: Anosmia; Hyposmia; Platelet-Rich Plasma (PRP); Intranasal Injection; Randomized Controlled Trial
MeSH Terms: conditions — Anosmia | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: Parallel two-arm design with participants randomly assigned to either carrier-assisted topical PRP application or intranasal PRP injection. Each participant receives only one type of intervention throughout the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and outcome assessors were blinded to the group assignment to minimize expectation bias. Interventions were prepared using an identical procedure to ensure blinding. The principal investigator, who was responsible for administering the intervention, was aware of group allocation. However, participants and outcome assessors had no access to allocation information throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal PRP injection (Experimental): Participants in this arm will receive an intranasal injection of autologous platelet-rich plasma (PRP) into the olfactory cleft. The procedure will be conducted under local anesthesia using endoscopic guidance. All participants will also perform standardized daily olfactory training for three months following the intervention.
  Interventions: Procedure: Intranasal Injection of Autologous PRP; Combination Product: platelet-rich plasma; Device: olfactory training
- Topical PRP application arm (Experimental): Participants in this arm will receive a topical application of autologous PRP delivered via PRP-soaked absorbable material (Gelfoam) placed into the olfactory cleft. No needle will be used. The placement will be guided by nasal endoscopy under local anesthesia. Daily olfactory training will be continued for three months post-application.
  Interventions: Procedure: Carrier-Assisted Topical Application of Autologous PRP; Combination Product: platelet-rich plasma; Device: olfactory training

INTERVENTIONS:
Procedure: Intranasal Injection of Autologous PRP — Under topical anesthesia and decongestion, approximately 1 mL of freshly prepared autologous platelet-rich plasma will be injected into multiple sites of the olfactory cleft mucosa bilaterally using a 25-gauge needle under endoscopic guidance. Single treatment session.
  Arms: Intranasal PRP injection
Procedure: Carrier-Assisted Topical Application of Autologous PRP — Four pieces of sterile, bioabsorbable carrier (Gelfoam sponge) will be soaked with approximately 5 mL of freshly prepared autologous platelet-rich plasma. Under endoscopic guidance, two pieces will be placed gently into each olfactory cleft, ensuring contact with the olfactory mucosa. Carriers will remain briefly to allow PRP diffusion before dissolving naturally or being removed. Single treatment session.
  Arms: Topical PRP application arm
Combination Product: platelet-rich plasma — This study adopts a fully automated, closed-system PRP preparation technique to ensure the stability of the blood product. A total of 60 mL of whole blood is drawn and processed using the Phoenix Q1 centrifuge (TFDA Medical Device Manufacturing License No. 004461) for blood component separation in a closed, sterile environment. An optical sensor identifies and automatically collects the buffy coat layer (rich in platelets and monocytes), yielding approximately 6 mL of autologous platelet-rich plasma (PRP). The centrifugation and PRP collection process takes about 5 minutes. Compared with traditional methods requiring manual identification and collection, this approach enhances the precision and safety of centrifugation-based preparation.
Device: olfactory training — Participants will perform olfactory training for 12 weeks following the PRP intervention. Training is conducted twice daily using four odor bottles containing standardized odorants from Sigma-Aldrich (Germany): lemon (citronellal, #27470), rose (phenylethanol, #77861), clove (eugenol, #W246700), and eucalyptus (eucalyptol, #C80601). Each odor is sniffed gently for about 20 seconds, with a 20-second pause between bottles. Participants will record the perceived intensity of each odor in a training diary after every session.

SUMMARY:
The goal of this clinical trial is to determine whether two different delivery methods of autologous platelet-rich plasma (PRP) can improve olfactory function in adults with persistent olfactory dysfunction lasting more than three months. The main questions it aims to answer are:

1. Does carrier-assisted topical application of PRP lead to comparable or better improvement in smell function than intranasal injection of PRP?
2. Which method provides greater patient comfort and fewer adverse effects?

Researchers will compare carrier-assisted topical PRP application to intranasal PRP injection to see if one approach is more effective in restoring olfactory function.

Participants will:

1. Receive a single PRP treatment delivered either by injection or via a PRP-soaked carrier placed into the olfactory cleft.
2. Continue daily olfactory training for three months following the intervention.
3. Undergo smell testing (Sniffin' Sticks) before and after treatment and complete quality-of-life questionnaires.

DETAILED DESCRIPTION:
Persistent olfactory dysfunction (OD) is a common sequela of viral upper respiratory tract infections, including COVID-19, and can significantly affect patients' quality of life, nutrition, and safety. Current treatment options are limited, with olfactory training being the primary evidence-based non-pharmacological therapy. Autologous platelet-rich plasma (PRP) is a concentration of platelets obtained from a patient's own blood, rich in growth factors and cytokines that promote neuronal regeneration, tissue repair, and neuroplasticity. Early clinical studies suggest PRP may improve olfactory function, but the optimal method for delivering PRP to the olfactory cleft remains unknown.

This randomized controlled trial will include a total of 60 adult patients aged 18-80 years old with olfactory loss (hyposmia or anosmia) persisting for more than 3 months despite standardized olfactory training, confirmed by a reduced Sniffin' Sticks TDI score.

PRP will be prepared on-site immediately before application using a standardized centrifugation protocol to achieve a platelet concentration 2-3 times above baseline. efficacy and safety of two PRP delivery methods will be compared:

Intranasal Injection Group: Autologous PRP will be injected directly into the mucosa of the olfactory cleft under endoscopic guidance. After topical anesthesia with lidocaine spray and decongestion with oxymetazoline, a 25-gauge needle will be used to deliver approximately 1 mL of PRP into multiple sites along the superior nasal cavity bilaterally.

Carrier-Assisted Topical Application Group: Four pieces of sterile, bioabsorbable carrier (Gelfoam sponge) will be soaked with approximately 5 mL of autologous PRP. Under endoscopic guidance, two pieces of PRP-soaked carrier will be placed gently into each side of olfactory cleft, ensuring contact with the olfactory mucosa. Carriers will remain in place for a short duration to allow diffusion of PRP before dissolving naturally or being removed.

Primary Outcome: Change in TDI score from baseline to 3 months post-treatment.

Secondary Outcomes: Patient-reported olfactory-related quality of life (QOD, SNOT-22, PQ), subjective improvement ratings, 20-item retronasal olfactory test, SSParoT, procedure tolerability, and adverse event rates.

Post-intervention care: All participants will continue standardized daily olfactory training for at least 12 weeks after PRP administration. Follow-up visits at 2 weeks, 1 month and 3 months will assess smell function, symptom changes, and safety.

This study aims to determine whether carrier-assisted topical PRP application is as effective or superior to intranasal PRP injection for improving olfactory function, while potentially offering a less invasive and more tolerable treatment approach. Results will help define optimal PRP delivery strategies for olfactory rehabilitation in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years, regardless of sex
* Subjective complaint of olfactory dysfunction with confirmed hyposmia or anosmia based on standardized olfactory testing
* History of at least 3 months of prior olfactory training but with persistent olfactory complaints

Exclusion Criteria:

* Congenital anosmia
* Diagnosed neurological or structural brain abnormalities (e.g., brain tumor, major head trauma, stroke) with low likelihood of olfactory recovery
* Inability or unwillingness to comply with study procedures or follow-up assessments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Sniffin' Sticks Olfactory Test | pre-intervention and at 1 and 3 months (may extend to 6 and 12 months) post-intervention
  The Sniffin' Sticks test (Burghart Messtechnik GmbH, Holm, Germany) comprises three subtests for odor detection threshold (T), odor discrimination (D), and odor identification (I). This test employs odor-containing felt-tip pens, which are presented to participants to evaluate their olfactory performance.
  In the detection threshold subtest, we employed an adaptive staircase procedure based on a three-alternative forced-choice format. Participants were tasked with differentiating a stick with a rose-like aroma (phenylethyl alcohol) from two blank sticks. Odor discrimination was assessed using 16 pen triplets, two of which contained identical odors and one stick contained a different odor. Participants were tasked with identifying the odd one out. In the odor identification subtest, participants were tasked with naming 16 common odors by selecting appropriate terms from a set of four descriptors per odor. The scores from each subtest were combined into a composite TDI score.

SECONDARY OUTCOMES:
Procedure-related pain evaluation | during the procedure and up to 2 weeks post-intervention
  Visual analogue scale for pain (0-10) immediately after procedure.
Retronasal Olfactory Test | pre-intervention and at 3 months post-intervention
  Retronasal olfactory testing was performed using standardized odorized powders/capsules presented in the oral cavity, with participants instructed to exhale through the nose and rate the perceived odor. It specifically evaluates olfactory function via the retronasal route.
Visual Analogus Scale for olfaction | pre-intervention and at 1 and 3 months (may extend to 6 and 12 months) post-intervention
  Visual Analogus Scale for olfactory function from 0 to 10. (0 means inability of smelling and 10 means super good smell function)
Questionnaire of Olfactory Disorders (QOD) | pre-intervention and at 1 and 3 months (may extend to 6 and 12 months) post-intervention
  A questionnaire on olfaction-related quality of life status
Beck Depression Inventory (BDI) | pre-intervention and 3 months post-intervention
  The Beck Depression Inventory (BDI) is a standardized self-report questionnaire measuring the severity of depressive symptoms. Olfactory loss, resulting from viral infections or other etiologies, has been associated with mood disturbances and reduced emotional well-being.
Montreal Cognitive Assessment (MoCA) | pre-intervention and post-3 month intervention
  The Montreal Cognitive Assessment (MoCA) is a widely used screening tool for mild cognitive impairment. Olfactory loss has been shown to diminish sensory stimulation to the brain, potentially affecting neural processing and cognitive function.
22-item Sinonasal Outcome Test (SNOT-22) | pre-intervention and at 1 and 3 months (may extend to 6 and 12 months) post-intervention
  A questionaire reflecting the severity of symptoms and the impact of sinonasal diseases
Parosmia Questionnaire (PQ) | pre-intervention and at 1 and 3 months (may extend to 6 and 12 months) post-intervention
  A 4-item questionnaire to evaluate the presence, severity, and qualitative characteristics of odor distortions (parosmia).
Sniffin' Sticks Parosmia Test | pre-intervention and 3 months post-intervention
  SSParoT (Sniffin' Sticks Parosmia Test) is a specialized assessment tool to evaluate qualitative olfactory function, particularly for the objective quantification of parosmia. It presents a series of well-characterized odorants and asks participants to rate each odor's pleasantness. From these ratings, the range of hedonic ratings and the hedonic orientation are calculated, providing quantitative measures of the breadth and direction of the participant's odor preference profile. This approach enables clinicians to identify patterns of altered odor perception and monitor changes following therapeutic interventions. The SSParoT (Sniffin' Sticks Parosmia Test) was additionally administered to participants with parosmia to calculate the range of hedonic ratings and the hedonic orientation.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding IPD sharing will be made upon completion of the study, pending institutional policies and ethical review board recommendations.

REFERENCES:
- [Background] Bae AY, Kim DH, Hwang SH. Efficacy of Platelet-Rich Plasma in the Treatment of Persistent Olfactory Impairment After COVID-19: A Systematic Review and Meta-Analysis. J Rhinol. 2024 Mar;31(1):1-7. doi: 10.18787/jr.2024.00006. Epub 2024 Mar 31. PMID 39664044
- [Background] Duffy A, Naimi B, Garvey E, Hunter S, Kumar A, Kahn C, Farquhar D, D'Souza G, Rawson N, Dalton P, Toskala E, Rabinowitz M, Rosen M, Nyquist G, Rosen D. Topical platelet-rich plasma as a possible treatment for olfactory dysfunction-A randomized controlled trial. Int Forum Allergy Rhinol. 2024 Sep;14(9):1455-1464. doi: 10.1002/alr.23363. Epub 2024 May 9. PMID 38722276
- [Background] Jiang RS, Chiang YF. The Effect of Platelet-Rich Plasma and Hyaluronic Acid Nasal Injections in the Treatment of Traumatic Olfactory Dysfunction. Ear Nose Throat J. 2024 Oct 15:1455613241291710. doi: 10.1177/01455613241291710. Online ahead of print. PMID 39404838
- [Background] Lechien JR, Le Bon SD, Saussez S. Platelet-rich plasma injection in the olfactory clefts of COVID-19 patients with long-term olfactory dysfunction. Eur Arch Otorhinolaryngol. 2023 May;280(5):2351-2358. doi: 10.1007/s00405-022-07788-8. Epub 2022 Dec 15. PMID 36520209
- [Background] Yan CH, Mundy DC, Patel ZM. The use of platelet-rich plasma in treatment of olfactory dysfunction: A pilot study. Laryngoscope Investig Otolaryngol. 2020 Feb 21;5(2):187-193. doi: 10.1002/lio2.357. eCollection 2020 Apr. PMID 32337347

DOCUMENTS (1):
  • Study Protocol (2025-07-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT07151703/Prot_000.pdf